CLINICAL TRIAL: NCT05038644
Title: MCW-XEN21: A Phase 1 Study of XmAb18968 (CD3-CD38) for the Treatment of Patients With Relapsed/Refractory CD38 Positive Acute Leukemia and T Cell Lymphoblastic Lymphoma
Brief Title: XmAb18968 (CD3-CD38) in Relapsed or Refractory Acute Leukemia and T Cell Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug expired May 31, 2024.
Sponsor: Ehab L Atallah (Other)
Responsible Party: Sponsor-Investigator, Ehab L Atallah, Professor, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO00041908
Record Dates: First submitted 2021-09-03; First posted 2021-09-09 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia; T Cell Acute Lymphoblastic Leukemia; T Cell Lymphoblastic Lymphoma
Keywords: XmAb18968
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Arm Z: Dose Level -1 for Group A (T-ALL, T-LBL) (Experimental): 0.1 mg intravenous (IV) Cycle (C) 1 Day (D) 1, 0.3 mg IV C1D2, then 0.4 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level -1
- Arm A: Dose Level 0 (Starting Dose) for Group A (T-ALL, T-LBL) (Experimental): 0.2 mg IV C1D1, 0.6 mg IV C1D2, then 0.8 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level 0 (starting dose)
- Arm B: Dose Level 1 for Group A (T-ALL, T-LBL) (Experimental): 0.25 mg IV C1D1, 0.75 mg IV C1D2, then 1.0 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level 1
- Arm C: Dose Level 2 Group A (T-ALL, T-LBL) (Experimental): 0.4 mg IV C1D1, 0.9 mg IV C1D2, then 1.3 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level 2
- Arm D: Dose Level 3 Group A (T-ALL, T-LBL) (Experimental): 0.5 mg IV C1D1, 1.0 mg IV C1D2, then 1.5 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level 3
- Arm Z: Dose Level -1 Group B (AML) (Experimental): 0.1 mg IV C1D1, 0.3 mg IV C1D2, then 0.4 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level -1
- Arm A: Dose Level 0 (Starting Dose) Group B (AML) (Experimental): 0.2 mg IV C1D1, 0.6 mg IV C1D2, then 0.8 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level 0 (starting dose)
- Arm B: Dose Level 1 Group B (AML) (Experimental): 0.25 mg IV C1D1, 0.75 mg IV C1D2, then 1.0 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level 1
- Arm C: Dose Level 2 Group B (AML) (Experimental): 0.4 mg IV C1D1, 0.9 mg IV C1D2, then 1.3 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level 2
- Arm D: Dose Level 3 Group B (AML) (Experimental): 0.5 mg IV C1D1, 1.0 mg IV C1D2, then 1.5 mg IV on D8, D15, and D22 in a 28-day cycle.
  Interventions: Drug: XmAb18968 - Dose level 3

INTERVENTIONS:
Drug: XmAb18968 - Dose level -1 — 0.1 mg IV C1D1, 0.3 mg IV C1D2, then 0.4 mg IV on D8, D15, and D22 in a 28-day cycle.
  Arms: Arm Z: Dose Level -1 Group B (AML); Arm Z: Dose Level -1 for Group A (T-ALL, T-LBL)
Drug: XmAb18968 - Dose level 0 (starting dose) — 0.2 mg IV C1D1, 0.6 mg IV C1D2, then 0.8 mg IV on D8, D15, and D22 in a 28-day cycle.
  Arms: Arm A: Dose Level 0 (Starting Dose) Group B (AML); Arm A: Dose Level 0 (Starting Dose) for Group A (T-ALL, T-LBL)
Drug: XmAb18968 - Dose level 1 — 0.25 mg IV C1D1, 0.75 mg IV C1D2, then 1.0 mg IV on D8, D15, and D22 in a 28-day cycle.
  Arms: Arm B: Dose Level 1 Group B (AML); Arm B: Dose Level 1 for Group A (T-ALL, T-LBL)
Drug: XmAb18968 - Dose level 2 — 0.4 mg IV C1D1, 0.9 mg IV C1D2, then 1.3 mg IV on D8, D15, and D22 in a 28-day cycle.
  Arms: Arm C: Dose Level 2 Group A (T-ALL, T-LBL); Arm C: Dose Level 2 Group B (AML)
Drug: XmAb18968 - Dose level 3 — 0.5 mg IV C1D1, 1.0 mg IV C1D2, then 1.5 mg IV on D8, D15, and D22 in a 28-day cycle.
  Arms: Arm D: Dose Level 3 Group A (T-ALL, T-LBL); Arm D: Dose Level 3 Group B (AML)

SUMMARY:
This is a phase 1, dose-escalation study (using 3 + 3 dose-limiting toxicity (DLT) criteria) evaluating the safety and tolerability of XmAb18968, as well as establishing a recommended phase II dose (RP2D) in subjects with T cell acute lymphoblastic leukemia (T-ALL) and T cell lymphoblastic (lymphoma) T-LBL (Group A) and acute myeloid leukemia (AML) (Group B).

DETAILED DESCRIPTION:
The primary objective of this portion of the study is to determine a recommended phase II dose (RP2D) for XmAb18968. The trial will use a variation of the 3 + 3 design where both escalation and de-escalation are possible. There will be separate cohorts; Group A (T cell acute lymphoblastic leukemia, T cell lymphoblastic lymphoma) and Group B (acute myeloid leukemia). A minimum of 24 and a maximum of 60 subjects will be needed for the study.

The first dose on Cycle 1 Day 1 (C1D1) will be split into two doses to ensure the safety of subjects and to closely monitor for CRS. The dose will be split into C1D1 and Cycle 1 Day 2 (C1D2) with approximately 25% of the dose given on C1D1 and 75% of the dose given on C1D2. Thereafter, subjects will receive the full dose planned for that cohort.

Prior to enrolling subjects at the next applicable dose level, the Data Safety Monitoring Committee (DSMC) will review the results.

Although AEs may occur at any point during treatment, only AEs occurring during Cycle 1 of treatment will necessarily influence decisions regarding dose escalation, expansion of a dose level, or evaluation of intermediate dose levels. Subjects will be monitored through all cycles of therapy for treatment-related toxicities.

Toxicity will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. If multiple AEs are seen, the presence of a DLT will be based on the most severe AE experienced. The DLT will be based on the tolerability observed during the first 28 days (or up to 42 days for hematological DLTs) of treatment/observation.

DLT will be defined as any of the following events:

* Any grade 4 or higher non-hematological adverse reaction.
* Cytokine release syndrome (CRS) is a possible side effect that can occur as a result of administration of XmAb18968. For this protocol, any grade 3 or higher CRS adverse event (AE) (per revised CRS grading system will be considered a DLT except grade 3 CRS AE that resolves to grade 1 within seven days).
* Any subject meeting the criteria for Hy's Law case (i.e., severe drug-induced liver injury (DILI)). A Hy's Law case is defined as: aspartate aminotransferase (AST) or alanine transaminase (ALT) values ≥ 3 × upper limit of normal (ULN) AND with serum total bilirubin (TBIL) level > 2 × ULN or international normalized ratio (INR) > 1.5 without signs of cholestasis.
* Any non-Hy's Law grade 3 liver abnormality lasting more than 72 hours will be considered a DLT.
* Grade 3 electrolyte abnormalities - sodium (Na), potassium (K), chloride (Cl), carbon dioxide (CO2), calcium (Ca), magnesium (Mg), phosphate - that do not return to grade 1 or lower within 72 hours.
* Any grade 4 neurotoxicity will be considered a DLT. Grade 3 neurotoxicity that lasts more than 72 hours will be considered a DLT.
* Any grade 3 nausea, vomiting, or diarrhea that requires hospitalization, tube feeding or total parenteral nutrition.
* Any adverse reaction that leads to dose reduction or withdrawal.
* Grade 3 transaminitis (AST/ALT) elevation that does not return to grade 1 or lower within 72 hours.
* Any grade 3 infection lasting more than seven days in the absence of active leukemia.
* Any grade 3 bleeding with thrombocytopenia in the absence of active leukemia.
* Any grade 4 or higher neutropenia lasting past cycle day 42 in the absence of active leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care.
2. Male or female subjects 18 years or older.
3. Morphologically documented T-ALL, AML (including undifferentiated leukemia and bi-phenotypic leukemia, or T-LBL in relapsed/refractory status (at least one line of prior therapy). Subjects with measurable residual disease by flow cytometry, molecular testing or cytogenetics will be eligible for the trial.
4. CD38 expression ≥ 20% by flow cytometry or immunohistochemistry at time of relapse.
5. Adequate organ system function as outlined below:

   1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN. If total bilirubin > 1.5 × ULN then check direct bilirubin. Subject will be eligible if direct bilirubin is < 1.5 × ULN.
   2. Calculated creatinine clearance ≥ 40 mL/min (calculated by Cockcroft-Gault formula) for subjects with creatinine levels above institutional normal.
   3. Ejection > 40% by echocardiogram or multiple-gated acquisition (MUGA) scan.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Female subjects who:

   1. Are postmenopausal for at least one year before the screening visit, OR
   2. Are surgically sterile, OR
   3. If they are of childbearing potential:

   i. Agree to practice one highly effective method and one additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through four months after the last dose of study drug (female and male condoms should not be used together), OR ii. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception).
8. Male subjects, even if surgically sterilized (i.e., status postvasectomy), who:

   1. Agree to practice effective barrier contraception during the entire study drug treatment period from the time of signing the informed consent through four months after the last dose of study drug (female and male condoms should not be used together), OR
   2. Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

Exclusion Criteria:

1. Acute promyelocytic leukemia.
2. Treatment with systemic antineoplastic therapy within 5 half-lives from the last dose before cycle one day one of therapy. Radiation within 7 days before C1D1 of therapy. The use of hydroxyurea, steroids, or vincristine for leukoreduction is permitted.
3. Prior treatment with an anti-CD38 antibody in last 6 months.
4. Hematopoietic stem cell transplantation within 6 months of enrollment, or evidence of veno-occlusive disease at any time post-transplant, or active graft-versus-host disease requiring immunosuppressive therapy.
5. Any serious medical or psychiatric illness that could, in the Investigator's opinion, potentially interfere with the completion of study procedures.
6. Active, significant, uncontrolled infection. Subjects with infections that are controlled by antibiotics, antiviral or antifungal therapy can be enrolled in the study.
7. Presence of another active malignancy (requiring treatment) treated within 12 months with the exception of:

   1. Adequately treated non-melanoma skin cancer,
   2. Adequately treated melanoma Grade 2 or less,
   3. Cervical intraepithelial neoplasia,
   4. Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast,
   5. Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin,
   6. Adequately treated prostate cancer.
8. Life-threatening illness with life expectancy < 6 months unrelated to cancer.
9. Subjects with active central nervous system (CNS) disease. Subjects with adequately treated CNS disease may enroll on the study.
10. Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection. Note: Subjects who have isolated positive hepatitis B core antibody (i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Subjects who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.
11. Known cardiopulmonary disease defined as:

    1. Unstable angina,
    2. Congestive heart failure (New York Heart Association [NYHA] Class III or IV;
    3. Myocardial infarction (MI) within six months prior to enrollment (subjects who had ischemic heart disease such as acute coronary syndrome, MI, and/or revascularization > 6 months before Screening and who are without cardiac symptoms may enroll),
    4. Clinically significant pulmonary hypertension requiring pharmacologic therapy,
    5. Clinically significant arrhythmia:

    i. History of polymorphic ventricular fibrillation or torsade de pointes, ii. Uncontrolled permanent atrial fibrillation (A-Fib), defined as continuous A-Fib for ≥ 6 months and not well controlled with adequate A-Fib therapy, iii. Uncontrolled persistent A-Fib, defined as sustained A-Fib lasting > 7 days and/or requiring cardioversion in the four weeks before Screening and not well controlled with A-Fib therapy, iv. Grade 3 A-Fib defined as symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation, and v. Subjects with paroxysmal A-Fib or < Grade 3 A-Fib for a period of at least 6 months are permitted to enroll provided that their rate is controlled on a stable regimen.
12. Subject has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, gastrointestinal or any other medical condition that in the opinion of the Investigator would adversely affect his/her participating in this study.
13. Uncontrolled high blood pressure as determined by the treating physician (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 100 mm Hg).
14. Subjects with uncontrolled coagulopathy or bleeding disorder.
15. Known moderate-to-severe chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis.
16. Major surgery within 14 days before the enrollment or a prescheduled major surgery during study period.
17. Female subjects who are both lactating and breastfeeding or of childbearing potential who have a positive serum or urine test during Screening.
18. Female subjects who intend to donate eggs (ova) during the course of this study or four months after receiving their last dose of study drug(s).
19. Male subjects who intend to donate sperm during the course of this study or four months after receiving their last dose of study drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
The number of dose-limiting toxicities for group A level -1 | 4 Years
  See DLT definitions in the detailed study description.
The number of dose-limiting toxicities for group A level 0 | 4 Years
  See DLT definitions in the detailed study description.
The number of dose-limiting toxicities for group A level 1 | 4 Years
  See DLT definitions in the detailed study description.
The number of dose-limiting toxicities for group A level 2 | 4 Years
  See DLT definitions in the detailed study description.
The number of dose-limiting toxicities for group A level 3 | 4 Years
  See DLT definitions in the detailed study description.
The number of dose-limiting toxicities for group B level -1 | 4 Years
  See DLT definitions in the detailed study description.
The number of dose-limiting toxicities for group B level 0 | 4 Years
  See DLT definitions in the detailed study description.
The number of dose-limiting toxicities for group B level 1 | 4 Years
  See DLT definitions in the detailed study description.
The number of dose-limiting toxicities for group B level 2 | 4 Years
  See DLT definitions in the detailed study description.
The number of dose-limiting toxicities for group B level 3 | 4 Years
  See DLT definitions in the detailed study description.
Recommended Phase 2 Dose for Group A | 4 Years
  This dose will be dependent on the number of dose-limiting toxicities reported in primary outcomes 1-5.
Recommended Phase 2 Dose for Group B | 4 Years
  This dose will be dependent on the number of dose-limiting toxicities reported in primary outcomes 6-10.

SECONDARY OUTCOMES:
The number of subjects with complete response in group A level -1. | 4 Years
  This is defined as no circulating lymphoblasts or extramedullary disease (no lymphadenopathy, splenomegaly). Testicular mass, skin/gum infiltration, CNS involvement; trilineage hematopoiesis with < 5% blasts; ANC > 1.0 × 10^9/L (1,000/μL); Platelet count > 100 × 10^9/L (100,000/μL); No recurrence for four weeks.
The number of subjects with complete response in group B level -1. | 4 Years
  This is defined as bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; ANC > 1.0 × 10^9/L (1,000/μL); platelet count > 100 × 10^9/L (100,000/μL); independence of red cell transfusions.
The number of subjects with complete response in group A level 0. | 4 Years
  This is defined as no circulating lymphoblasts or extramedullary disease (no lymphadenopathy, splenomegaly). Testicular mass, skin/gum infiltration, CNS involvement; trilineage hematopoiesis with < 5% blasts; ANC > 1.0 × 10^9/L (1,000/μL); Platelet count > 100 × 10^9/L (100,000/μL); No recurrence for four weeks.
The number of subjects with complete response in group B level 0. | 4 Years
  This is defined as bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; ANC > 1.0 × 10^9/L (1,000/μL); platelet count > 100 × 10^9/L (100,000/μL); independence of red cell transfusions.
The number of subjects with complete response in group A level 1. | 4 Years
  This is defined as no circulating lymphoblasts or extramedullary disease (no lymphadenopathy, splenomegaly). Testicular mass, skin/gum infiltration, CNS involvement; trilineage hematopoiesis with < 5% blasts; ANC > 1.0 × 10^9/L (1,000/μL); Platelet count > 100 × 10^9/L (100,000/μL); No recurrence for four weeks.
The number of subjects with complete response in group B level 1. | 4 Years
  This is defined as bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; ANC > 1.0 × 10^9/L (1,000/μL); platelet count > 100 × 10^9/L (100,000/μL); independence of red cell transfusions.
The number of subjects with complete response in group A level 2. | 4 Years
  This is defined as no circulating lymphoblasts or extramedullary disease (no lymphadenopathy, splenomegaly). Testicular mass, skin/gum infiltration, CNS involvement; trilineage hematopoiesis with < 5% blasts; ANC > 1.0 × 10^9/L (1,000/μL); Platelet count > 100 × 10^9/L (100,000/μL); No recurrence for four weeks.
The number of subjects with complete response in group B level 2. | 4 Years
  This is defined as bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; ANC > 1.0 × 10^9/L (1,000/μL); platelet count > 100 × 10^9/L (100,000/μL); independence of red cell transfusions.
The number of subjects with complete response in group A level 3. | 4 Years
  This is defined as no circulating lymphoblasts or extramedullary disease (no lymphadenopathy, splenomegaly). Testicular mass, skin/gum infiltration, CNS involvement; trilineage hematopoiesis with < 5% blasts; ANC > 1.0 × 10^9/L (1,000/μL); Platelet count > 100 × 10^9/L (100,000/μL); No recurrence for four weeks.
The number of subjects with complete response with incomplete hematological recovery in group A level -1. | 4 Years
  Meets all criteria for CR except absolute neutrophil count (ANC) or platelet count.
The number of subjects with complete response with incomplete hematological recovery in group B level -1. | 4 Years
  All complete response (CR criteria) except for residual neutropenia (< 1.0 × 10^9/L [1,000/μL]) or thrombocytopenia (< 100 × 10^9/L [100,000/μL]).
The number of subjects with complete response with incomplete hematological recovery in group A level 0 (starting dose). | 4 Years
  Meets all criteria for CR except absolute neutrophil count (ANC) or platelet count.
The number of subjects with complete response with incomplete hematological recovery in group B level 0 (starting dose). | 4 Years
  All complete response (CR criteria) except for residual neutropenia (< 1.0 × 109/L [1,000/μL]) or thrombocytopenia (< 100 × 109/L [100,000/μL]).
The number of subjects with complete response with incomplete hematological recovery in group A level 1. | 4 Years
  Meets all criteria for CR except absolute neutrophil count (ANC) or platelet count.
The number of subjects with complete response with incomplete hematological recovery in group B level 1. | 4 Years
  All complete response (CR criteria) except for residual neutropenia (< 1.0 × 109/L [1,000/μL]) or thrombocytopenia (< 100 × 109/L [100,000/μL]).
The number of subjects with complete response with incomplete hematological recovery in group A level 2. | 4 Years
  Meets all criteria for CR except absolute neutrophil count (ANC) or platelet count.
The number of subjects with complete response with incomplete hematological recovery in group B level 2. | 4 Years
  All CR criteria except for residual neutropenia (< 1.0 × 109/L [1,000/μL]) or thrombocytopenia (< 100 × 109/L [100,000/μL]).
The number of subjects with complete response with incomplete hematological recovery in group A level 3. | 4 Years
  Meets all criteria for CR except ANC or platelet count.
The number of subjects with complete response with incomplete hematological recovery in group B level 3. | 4 Years
  All complete response (CR criteria) except for residual neutropenia (< 1.0 × 109/L [1,000/μL]) or thrombocytopenia (< 100 × 109/L [100,000/μL]).
Event-free survival (EFS) in group A | 4 Years
  EFS will be defined from the time of achievement of CR/CRi to the time of next relapse/progression/death as measured by the National Comprehensive Cancer Network (NCCN) Response Criteria for Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma.
Event-free survival (EFS) in group B | 4 Years
  EFS will be will be defined from the time of achievement of CR/CRi to the time of next relapse/progression/death as measured by the Response Evaluation Criteria: Acute Myeloid Leukemia.
Overall survival in group A | 4 Years
  The length of time from when a subject begins treatment until death due to any cause.
Overall survival in group B. | 4 Years
  The length of time from when a subject begins treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Atallah, MD, Principal Investigator — Medical College of Wisconsin
Locations (6):
- United States (6):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Oregon Health & Science University, Portland, Oregon
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No